CLINICAL TRIAL: NCT03524963
Title: A Randomized, Open Label, Multiple Does, Crossover Study to Compare the Safety/Tolerability and Pharmacokinetics Between Pleetal SR Cap. and Cilostan CR Tab. in Healthy Volunteers
Brief Title: Comparative Pharmacokinetic Study Between Two Extended-Release Cilostazol Formulations in Korea
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bundang CHA Hospital (Other)
Responsible Party: Principal Investigator, Doo-Yeoun Cho, M.D., Professor, Bundang CHA Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 021-402-00016
Record Dates: First submitted 2018-05-01; First posted 2018-05-15 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Experimental): Cilostan CR Tab. in phase 1 and Pletaal SR Cap. in phase 2
  Interventions: Drug: Cilostan CR Tab.; Drug: Pletaal SR Cap.
- Sequence B (Experimental): Pletaal SR Cap. in phase 1 and Cilostan CR Tab. in phase 2
  Interventions: Drug: Cilostan CR Tab.; Drug: Pletaal SR Cap.

INTERVENTIONS:
Drug: Cilostan CR Tab. — Cilostan CR Tab. 200mg once a day for 5 days
Drug: Pletaal SR Cap. — Pletaal SR Cap. 200mg once a day for 5 days

SUMMARY:
This is a randomized, open-label, multiple-dose, two-sequence, two-period crossover study to to compare the safety/tolerability and pharmacokinetics between Pletaal SR Cap. and Cilostan CR Tab. in healthy volunteers

DETAILED DESCRIPTION:
Eligibility for participation of this study will be determined from demographic information, medical history, physical examination, electrocardiogram (ECG) and clinical laboratory tests within 4 weeks before study drug administration. Subjects suitable for this study will be admitted to the Clinical Trial Center of CHA Bundang Medical Center on the day before dosing (Day -1).

From Day 1 to 5, Subjects will be dosed study drug (Pletaal SR Cap. 200 mg once a day or Cilostan CR Tab. 200mg once a day).

Pharmacokinetic samplings will be done upto 24 hours after 1st study drug dosing and upto 72 hours after 5th study drug dosing.

After 9 days of washout period (Day 15), Subjects will be dosed study drug and pharmacokinetic samplings will be done by crossover manner.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects aged 20 - 45 years
* BMI (body mass index) between 18.0 and 27.0
* Agreement with written informed consent

Exclusion Criteria:

* Clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal disease or mental disorder (Past history or present)
* Inadequate result of laboratory test (especially, ALT/AST/r-GTP/ALP/LDH/Total bilirubin > 1.5 x UNL)
* Positive reaction in the HBs Ag, anti-HCV Ab, anti-HIV Ab
* Taking OTC (Over the counter) medicine including oriental medicine within 7 days
* Clinically significant allergic disease
* Subject with known for hypersensitivity reaction to Cilostazol
* Previous whole blood donation within 60 days or component blood donation within 30 days
* Previous participation of other trial within 90 days
* Continued taking caffeine (caffeine > 5 cup/day), drinking (alcohol > 30 g/day) and severe heavy smoker (cigarette > 1/2 pack per day)

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Cmax | up to 24 hours after 1st dose
  Maximal plasma concentration
AUC0-24 | up to 24 hours after 1st dose
  Area under the time-concentration curve
Cmax,ss | up to 72 hours after 5th dose
  Maximal plasma concentration at steady-state
AUCtau | up to 24 hours after 5th dose
  Area under the time-concentration curve

SECONDARY OUTCOMES:
AE | Up to 30 days after final dose
  Adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- CHA Bundang Medical Center, Seongnam, South Korea

IPD SHARING:
Plan to Share IPD: Undecided